CLINICAL TRIAL: NCT04702178
Title: A Randomized, Observer-Blind, Dose-Escalation Phase 1 Clinical Trial of COVAC-2 in Healthy Adults
Brief Title: A Clinical Trial of COVAC-2 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Government of Canada (Other Government); Government of Saskatchewan (Other Government); Vaccine Formulation Institute (VFI) (Unknown); Seppic (Industry)
Responsible Party: Principal Investigator, Volker Gerdts, Director & CEO Vaccine and Infectious Disease Organization, University of Saskatchewan
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVAC-001
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: interventions — COVAC-1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Group A-2 (Experimental): COVAC-2 25 µg: 8 healthy adults 18 to 54 years of age receive the vaccine on Day 0, followed by a second dose on Day 28.
  Interventions: Biological: COVAC-2
- Group B-2 (Placebo Comparator): Placebo Control: 4 healthy adults 18 to 54 years of age receive a dose of normal saline (placebo) on Day 0, followed by a dose of normal saline (placebo) on Day 28.
  Interventions: Biological: Saline Placebo
- Group C-2 (Experimental): COVAC-2 50 µg: 8 healthy adults 18 to 54 years of age receive the vaccine on Day 0, followed by a second dose on Day 28.
  Interventions: Biological: COVAC-2
- Group D-2 (Placebo Comparator): Placebo Control: 4 healthy adults 18 to 54 years of age receive a dose of normal saline (placebo) on Day 0, followed by a dose of saline placebo on Day 28.
  Interventions: Biological: Saline Placebo
- Group E-2 (Experimental): COVAC-2 100 µg: 8 healthy adults 18 to 54 years of age receive the vaccine on Day 0, followed by a second dose on Day 28.
  Interventions: Biological: COVAC-2
- Group F-2 (Placebo Comparator): Placebo Control: 4 healthy adults 18 to 54 years of age receive a dose of normal saline (placebo) on Day 0, followed by a dose of saline placebo on Day 28.
  Interventions: Biological: Saline Placebo
- Group G-2 (Experimental): COVAC-2 25 µg: 8 or 9 healthy adults ≥ 55 years of age receive the vaccine on Day 0, followed by a second dose on Day 28.
  Interventions: Biological: COVAC-2
- Group H-2 (Placebo Comparator): Placebo Control: 4 or 5 healthy adults ≥ 55 years of age receive a dose of normal saline (placebo) on Day 0, followed by a dose of normal saline (placebo) on Day 28.
  Interventions: Biological: Saline Placebo
- Group I-2 (Experimental): COVAC-2 50 µg: 8 healthy adults ≥ 55 years of age receive the vaccine on Day 0, followed by a second dose on Day 28.
  Interventions: Biological: COVAC-2
- Group J-2 (Placebo Comparator): Placebo Control: 4 healthy adults ≥ 55 years of age receive a dose of normal saline (placebo) on Day 0, followed by a dose of saline placebo on Day 28.
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: COVAC-2 — Intramuscular vaccine against SARS-CoV-2
  Arms: Group A-2; Group C-2; Group E-2; Group G-2; Group I-2
Biological: Saline Placebo — Intramuscular injection of saline placebo
  Arms: Group B-2; Group D-2; Group F-2; Group H-2; Group J-2

SUMMARY:
VIDO has developed a vaccine called COVAC-2.

The study vaccine contains a portion of the SARS-CoV-2 spike protein, called S1. The spike protein is the part of the virus that is responsible for attaching to the surface of host cells. COVAC-2 contains a SWE adjuvant. An adjuvant is a compound that is added to a vaccine to help the vaccine produce a better immune response. The SWE adjuvant belongs to a family of oil-based adjuvants that have been given to millions of people around the world as part of influenza vaccines. The COVAC-2 vaccine is expected to stimulate the body to make antibodies against the S1 protein. The antibodies will recognize the viral spike protein if the body is exposed to the virus and prevent or reduce the severity of COVID-19 illness. In animal studies, the immune response generated by the COVAC-2 vaccine was able to protect the vaccinated animals against a severe SARS-CoV-2 infection.

Phase 1 is a multi-centred trial of the COVAC-2 vaccine to be completed in Canada. It will be a randomized, observer-blinded, and placebo-controlled study to assess the safety and immunogenicity of three dosing levels (25, 50, and 100 µg protein) administered twice (4 weeks apart) in healthy adults 18 through 54 years of age (Phase 1a) and 55 years of age and older (Phase 1b).

Enrolment and vaccination of participants will be staggered over time based on participant age and vaccine dose. Approval will be sought from the Data Safety Monitoring Board (DSMB) to proceed with the second dose in each group, to enroll at each dose level, and to enroll in the older age group for each dose level.

Within the same age group, the 8 participants receiving the lowest dose are randomized with 4 participants receiving placebo; the 8 participants receiving the medium dose are randomized with 4 participants receiving placebo; and the 8 participants receiving the highest dose are randomized with 4 participants receiving placebo.

Within each dose level of 12 participants, it is proposed to immunize a first cohort of 3 participants (including at least 2 active vaccine participants) and pending no holding rule is met after 48 hours, to immunize the remaining 9 participants within that dose level.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy all of the following criteria:

1. Male and female healthy adults ages 18 years of age or older;
2. Good general health as determined by screening evaluation no greater than 30 days before immunization;
3. If female of child-bearing potential and heterosexually active, practice of adequate contraception for 30 days prior to injection, negative pregnancy test on the day of injection, and agreement to continue adequate contraception until 180 days after the second injection and;
4. Written informed consent, after review of the consent form and having adequate opportunity to discuss the study with an investigator or a qualified designee.

Exclusion Criteria:

Participant with any of the following criteria will be excluded:

1. Presence of any febrile illness or any known or suspected acute illness on the day of any immunization;
2. Any physical findings suggestive of acute or chronic illness;
3. Any immunodeficiency (congenital or acquired);
4. Receiving systemic immunosuppressive therapy or history of receiving chemotherapy in last 5 years other than topical agents;
5. Receipt of systemic glucocorticoids (a dose ≥ 20 mg/day prednisone or equivalent for 14 days) within 1 month, or any other cytotoxic or immunosuppressive drug within 6 months;
6. Cancer diagnosis in the last 5 years, excluding basal cell and squamous cell carcinoma of the skin, which are allowed;
7. Presence of autoimmune disease;
8. Receipt of any investigational drug within 6 months;
9. Receipt of any non-COVID-19 authorized vaccines within 2 weeks of study immunization;
10. Receipt of any authorized COVID-19 vaccine prior to study enrollment;
11. Receipt of any other experimental SARS-CoV-2/COVID-19 or other experimental coronavirus vaccine(s) at any time prior to or during the study;
12. Receipt of blood products or immunoglobulin (IVIg or IMIg) within 3 months of study entry/baseline serologic evaluation;
13. Current anti-tuberculosis therapy;
14. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine;
15. Hematologic or biochemical laboratory abnormalities (blood or urine), as defined by lab normal ranges. To exclude transient abnormalities, the investigator may repeat a test once, and if the repeat test is normal according to local reference ranges, participant may be enrolled. Grade 1 abnormalities of laboratory values will not be exclusionary if considered not clinically significant by the investigator and;
16. Known current or previous laboratory-confirmed SARS-CoV-1 OR SARS-CoV-2 infection, as documented by a positive polymerase chain reaction (PCR) test from a nasal swab OR known or laboratory-confirmed positive serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) from the first injection to Day 28, in all participants, in all groups | Day 0 - 28
  * The occurrence of each solicited local and general AE, during each 7-day follow-up period after injection (e.g. the day of injection and 6 subsequent days);
  * The occurrence of any unsolicited AEs for the entire study period;
  * The occurrence of any hematological (hemoglobin level, WBC, lymphocyte, neutrophil, eosinophil, and platelet count) and biochemical (ALT, AST, BUN, and Cr) clinically significant laboratory abnormality through to Day 28 and;
  * The occurrence of any serious AEs (SAEs), medically attended events (MAE), or adverse event of special interest (AESI).
Occurrence of AEs from the second injection to Day 56 (28 days post injection), in all participants, in all groups | Day 28 - 56
  * The occurrence of solicited local and general AE, during each 7-day follow-up period after the second injection (e.g. the day of 2nd injection and 6 subsequent days);
  * The occurrence of any unsolicited AEs for the entire study period

SECONDARY OUTCOMES:
Specific antibody response induced by the vaccine against the SARS-CoV-2 S protein as measured by ELISA | Days 0, 7, 14, 28, 35, 42, 56, 90, 120, and 365
  The immune response to the study vaccine, as measured by antibody (e.g. IgG and other isotypes) directed to Wuhan spike antigen or neutralizing antibodies pre-injection (Day 0) and post-injection(s)
Specific cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus | Days 0, 14, 28, 35, 42, 120, and 365
  o The immune response to the study vaccine, as measured by cell immune response markers in PBMCs collected pre-injection (Day 0) and post-injection(s)

OTHER OUTCOMES:
Specific antibody response induced by the vaccine against the SARS-CoV-2 RBD protein as measured by ELISA | Days 0, 7, 14, 28, 35, 42, 56, 90, 120, and 365
  • The immune response to the study vaccine, as measured by antibody directed to RBD antigen pre-injection (Day 0) and post-injection(s)
Specific neutralizing antibody response induced by the vaccine against the B.1.1.7 Variant of Concern, as measured by neutralization assay. | Days 0, 7, 14, 28, 35, 42, 56, 90, 120, and 365
  The immune response to the study vaccine, as measured by neutralizing antibodies against Variant of Concern B.1.1.7 pre-injection (Day 0) and post-injection(s).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Langley, MD, Principal Investigator — Canadian Center for Vaccinology
Locations (2):
- Canada (2):
  - Canadian Center for Vaccinology, Dalhousie University, Halifax, Nova Scotia
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garg R, Liu Q, Van Kessel J, Asavajaru A, Uhlemann EM, Joessel M, Hamonic G, Khatooni Z, Kroeker A, Lew J, Scruten E, Pennington P, Deck W, Prysliak T, Nickol M, Apel F, Courant T, Kelvin AA, Van Kessel A, Collin N, Gerdts V, Koster W, Falzarano D, Racine T, Banerjee A. Efficacy of a stable broadly protective subunit vaccine platform against SARS-CoV-2 variants of concern. Vaccine. 2024 Aug 13;42(20):125980. doi: 10.1016/j.vaccine.2024.05.028. Epub 2024 May 19. PMID 38769033